CLINICAL TRIAL: NCT03163849
Title: Assessment of Haematological and Biochemical Effect After New Direct Acting Antiviral Drugs in Chronic Hepatitis c Virus Egyptian Patients in Assiut Province
Brief Title: Assessment Effects After Direct Acting Antiviral in Chronic Hepatitis c Virus Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sahar Ezeldeen Hussein Ali, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRHCV
Record Dates: First submitted 2017-05-18; First posted 2017-05-23 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): oral tablets
  Interventions: Drug: Placebos
- Study group (Experimental): sofosbuvir , daclatasvir oral tablets
  Interventions: Drug: Sofosbuvir , daclatasvir

INTERVENTIONS:
Drug: Sofosbuvir , daclatasvir — Tablets
  Arms: Study group
Drug: Placebos — oral tablets
  Arms: control group

SUMMARY:
Chronic hepatitis C virus infection affects an estimated one hundred and seventy million people around the world with and approximate prevalence 0.2-2 % in the United State of America and European countries.

DETAILED DESCRIPTION:
In Egypt, Chronic hepatitis C virus is a serious health problem where Chronic hepatitis C virus prevalence is very high.

Chronic Chronic hepatitis C virus infection is associated with a high risk for liver-related mortality because of a variety of complications, which appear obviously in those patients with developing end-stage liver disease, including decompensated liver cirrhosis and hepatocellular carcinoma. Egypt had the highest burden of deaths from Chronic hepatitis C virus-associated hepatocellular carcinoma in the Arab world, around sixty three percentage of all Chronic hepatitis C virus-associated hepatocellular carcinoma deaths happened in Egypt.

Poor response rates and poor tolerability were observed during treatment of chronic Chronic hepatitis C virus infection with pegylated interferon and ribavirin.

Because Chronic hepatitis C virus does not incorporate into the human genome and must replicate to maintain infection, it should be potential to destroy the virus completely by blocking replication at one or more stages of the life cycle.

In recent years, there has been a shift in treatment paradigm with the discovery and approval of agents that target specific proteins vital for hepatitis C replication. The Non Structural 3/4A inhibitors simeprevir and paritaprevir, the NonStructural 5A inhibitors ombitasvir, ledipasvir, and daclatasvir, and the Non Structural 5B inhibitors sofosbuvir and dasabuvir have been approved and incorporated as first-line agents into the latest guidelines for Hepatitis C treatment. Used in combination, these agents produce higher rates of sustained virologic response and less adverse effects than historical options, along with limited rates of resistance.

In previous studies ,haematological side effect of interferon and Ribavirin was reported in the form of reduction in Haemoglobin ,White Blood Cells and asymptomatic thrombocytopenia While SOF based combination therapy improved the liver function, anemia ,leucopenia and thrombocytopenia were detected especially after treatment with SOF,RBV and PegINF alpha .also significant improvement in the level of ALT and AST post treatment with either SOF and RBV or SOF ,RBV and INF were detected as compaired to baseline While no significant differences were detected on the level of total bilirubin or creatinine In our study we will assess and evaluate many biochemical and hematological findings upon new direct acting antiviral agents in Egyptian chronic hepatitis C virus patients

ELIGIBILITY:
Inclusion Criteria:

* Our study proposed for all consented patients complaining from chronic Hepatitis C virus infection undergoing treatment with antiviral drugs is possible through certain indications or criteria as follow:
* Patients with chronic Hepatitis C virus who are candidates for Direct Acting Antiviral Therapy:
* Age is from 18 to 65 years.

Exclusion Criteria:

* Those patients with chronic Hepatitis C virus infection are impossible or contraindicated to be treated with antiviral drugs as follow: - Geriatrics (> 65 years of age): - Pediatrics (< 18 years of age): - patients with known hypersensitivity to any of the components of the antiviral drug.
* Post-Liver Transplant Patients. ـPatients with primary haematological abnormalities not related to chronic hepatitis C virus infection
* Experienced patients (previously failed treatment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients with hematological changes | 12 weeks
  complete blood count and prothrombin time and concentration
The percentage of patients with antibodies against RBCs | Pre treatment
  Coomb's test

SECONDARY OUTCOMES:
the percentage of patients with biochemical changes | 12 weeks
  Urea, creatinine,bilirubin,ALT,AST
The percentage of patients with antibodies against RBCs | Three months after the end of treatment
  Coomb's test

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Ali, Master Degree, Principal Investigator — Internal medicine
Locations (2):
- Egypt (2):
  - Assuit, Asyut, Assuit
  - Assuit, Asyut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esteban JI, Sauleda S, Quer J. The changing epidemiology of hepatitis C virus infection in Europe. J Hepatol. 2008 Jan;48(1):148-62. doi: 10.1016/j.jhep.2007.07.033. Epub 2007 Nov 5. PMID 18022726
- [Background] Lavanchy D. The global burden of hepatitis C. Liver Int. 2009 Jan;29 Suppl 1:74-81. doi: 10.1111/j.1478-3231.2008.01934.x. PMID 19207969
- [Background] Darwish NM, Abbas MO, Abdelfattah FM, Darwish MA. Hepatitis C virus infection in blood donors in Egypt. J Egypt Public Health Assoc. 1992;67(3-4):223-36. PMID 1296960
- [Background] Fallahian F, Najafi A. Epidemiology of hepatitis C in the Middle East. Saudi J Kidney Dis Transpl. 2011 Jan;22(1):1-9. PMID 21196607
- [Background] El-Serag HB, Mason AC. Rising incidence of hepatocellular carcinoma in the United States. N Engl J Med. 1999 Mar 11;340(10):745-50. doi: 10.1056/NEJM199903113401001. PMID 10072408
- [Background] Davis GL, Albright JE, Cook SF, Rosenberg DM. Projecting future complications of chronic hepatitis C in the United States. Liver Transpl. 2003 Apr;9(4):331-8. doi: 10.1053/jlts.2003.50073. PMID 12682882
- [Background] Verna EC, Brown RS Jr. Hepatitis C virus and liver transplantation. Clin Liver Dis. 2006 Nov;10(4):919-40. doi: 10.1016/j.cld.2006.08.012. PMID 17164125
- [Background] Khan G, Hashim MJ. Burden of virus-associated liver cancer in the Arab world, 1990-2010. Asian Pac J Cancer Prev. 2015;16(1):265-70. doi: 10.7314/apjcp.2015.16.1.265. PMID 25640363
- [Background] Operskalski EA, Kovacs A. HIV/HCV co-infection: pathogenesis, clinical complications, treatment, and new therapeutic technologies. Curr HIV/AIDS Rep. 2011 Mar;8(1):12-22. doi: 10.1007/s11904-010-0071-3. PMID 21221855
- [Background] Chayama K, Hayes CN. HCV Drug Resistance Challenges in Japan: The Role of Pre-Existing Variants and Emerging Resistant Strains in Direct Acting Antiviral Therapy. Viruses. 2015 Oct 13;7(10):5328-42. doi: 10.3390/v7102876. PMID 26473914